CLINICAL TRIAL: NCT03649230
Title: A Phase IV, Real World Observational Study On The Use Of Akynzeo® (Netupitant/Palonosetron) For The Prevention Of Nausea and Vomiting in Oncology Patients Receiving Highly Emetogenic Chemotherapy (HEC) Over Multiple Cycles.
Brief Title: Observational Study on the Use of Akynzeo® in Patients Receiving HEC
Acronym: EVOLVE_CINV
Status: Completed | Type: Observational
Sponsor: Purdue Pharma, Canada (Industry)
Responsible Party: Sponsor
Other Study IDs: CAN-PRO-NEPA-001
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2022-10

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — netupitant, palosentron drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: 300mg netupitant/0.5mg palonosetron hydrochloride — Antiemetic (NK1 receptor antagonist/5-HT3 receptor antagonist)
  Other Names: Akynzeo®

SUMMARY:
This Canadian, multi-centre, prospective, observational real-world study is designed to collect patient-reported outcome data on the use of Akynzeo® (netupitant/palonosetron) for the prevention of nausea and vomiting in oncology patients receiving highly emetogenic chemotherapy (HEC).

DETAILED DESCRIPTION:
The study will assess quality of life using the Functional Living Index of Emesis (FLIE) questionnaire and generate Real World Evidence in support of existing clinical trial data, including effectiveness and safety of Akynzeo® in the real world setting for the prevention of Chemotherapy Induced Nausea and Vomiting (CINV) in patients receiving highly emetogenic chemotherapy (HEC).

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Patient scheduled to receive a highly emetogenic chemotherapy (HEC).
2. Patient scheduled to receive antiemetic prevention with Akynzeo® according to the approved Canadian Product Monograph as deemed medically necessary by the participating physician independently from this study.
3. Age ≥ 18 years.
4. Women of childbearing potential must use effective contraception during therapy and up to one month after treatment with Akynzeo®.
5. Patient (and/or patient's authorized legal representative) should understand the nature of the study and provide written informed consent prior to or at the screening visit.
6. Patient is able and willing to comply with the study protocol for the entire length of the study and will follow all study requirements, procedures and complete all visits as required.
7. Patient is participating in another clinical trial where antiemetic treatment is not pre-specified by the study protocol.

Exclusion Criteria:

1. Women of child bearing potential who are pregnant, planning on becoming pregnant or breast feeding.
2. Hypersensitivity to active substances, excipients or other ingredients of Akynzeo®.
3. Concomitant use of pimozide, terfenadine, astemizole, or cisapride.
4. Patient currently enrolled in another clinical trial where antiemetic treatment is pre-specified by the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult male or female chemotherapy patients of various cancer types who are scheduled to receive chemotherapy with high emetogenic potential for a maximum of 2 days.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jodan Ratz, PhD, Study Director — Purdue Pharma, Canada
Locations (17):
- Canada (17):
  - Tom Baker Cancer Center, Calgary, Alberta
  - The Moncton Hospital, Moncton, New Brunswick
  - NSHA-QEII Health Sciences Centre, Halifax, Nova Scotia
  - Cape Breton Cancer Centre, Sydney, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - William Osler Health System, Brampton, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Centre Integre de Sante et de Services Sociaux de la Monteregie-Centre, Greenfield Park, Quebec
  - Cisss de Chaudiere-Appalaches, Lévis, Quebec
  - Segal Cancer Centre-Jewish General Hospital, Montreal, Quebec
  - Centre de recherche du CHUS and Hopital Fleurimont, Sherbrooke, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from cancer treatment centers based on physician review of medical charts from the recruiting physicians clinical practice and referral from other physicians.
Groups:
- Treatment: 300mg netupitant/0.5mg palonosetron hydrochloride
Period: Overall Study
Arm/Group | Treatment
Started | 207
Completed | 150
Not Completed | 57
Not completed — Adverse Event | 12
Not completed — Death | 8
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 5
Not completed — Disease progression | 5
Not completed — Switched to non-HEC | 5
Not completed — Chemotherapy discontinued | 4
Not completed — Received only 3 HEC cycles | 4
Not completed — Screen Failure | 3
Not completed — Patient stopped treatment | 2
Not completed — Protocol Violation | 1
Not completed — Non-compliance | 1
Not completed — Patient Received Cisplatin days 1-3 q 3 weeks | 1

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat population includes all patients who were included in the ITT population and fulfilled all entry criteria and received at least one dose of the study treatment. 10 patients in the ITT population did not receive at least one dose of the study treatment.
Groups:
- Modified Intent-to-Treat Population: 300mg netupitant/0.5mg palonosetron hydrochloride
Arm/Group | Modified Intent-to-Treat Population
Number analyzed (Participants) | 197
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.0 [50.0 to 68.0]
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean (SD) | 58.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161
  Male | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 168
  Hispanic | 2
  Black | 6
  Aboriginal | 2
  Asian | 14
  other | 5
Region of Enrollment [Count of Participants; unit: Participants] — This study was only conducted in Canada.
  Participants
    Canada | 197

OUTCOME MEASURES:

1. Primary Outcome: Total Functional Living Index-Emesis (FLIE) Score at Cycle 1
Description: The Functional Living Index - Emesis questionnaire is a validated patient reported outcome with the objective of assessing the impact of chemotherapy-induced nausea and vomiting on patient's daily function.
  Questionnaire consists of a nausea domain and a vomiting domain of nine items each where the patient should rate how much nausea and vomiting have affected the quality of life. For each question the patient will rate how much nausea (or vomiting) has affected an aspect of his quality of life during the past five days. Each question uses a visual analogue scale (100 mm) and an ordinal scale (where 1= no emesis-7=a great deal). The minimum total score is 18 and the maximum total score is 126. Higher scores indicate less impairment on daily life as a result of nausea or vomiting. A FLIE total score > 108 indicates no impairment on daily life as a result of nausea or vomiting.
  Assessed by patient following day 5 of each cycle.
Time Frame: Day 5 of cycle 1
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 184
score on a scale | 109.2 (17.7)

2. Secondary Outcome: Complete Response
Description: No emetic episode and no use of rescue medication in the overall period (0-120h/Day 1-5)
Time Frame: Days 1-5 (0 - 120 hours) of cycles 1, 2, 3, 4; each cycle is approximately 28 days
Population: mITT
Measure: Count of Participants; unit: Participants
Groups:
- Cycle 1; Cycle 2; Cycle 3; Cycle 4: 300mg netupitant/0.5mg palonosetron hydrochloride
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3 | Cycle 4
Number analyzed (Participants) | 196 | 184 | 175 | 151
Participants
  Complete Response: Yes | 84 | 97 | 104 | 101
  Complete Response: No | 96 | 78 | 62 | 44
  Missing Data | 16 | 9 | 9 | 6

3. Secondary Outcome: Severity of Nausea on Day 5 (Change From Day 1)
Description: Question 1 of the daily evaluation of the Patient Diary ("How much nausea did you experience on average during the last 24 hours?"). Data was collected on a visual analogue scale. Scale ranges from 0 mm ("no nausea") to 100 mm ("always severe nausea").
Time Frame: Days 1-5 (0 - 120 hours) of cycles 1, 2, 3, 4; each cycle is approximately 28 days
Population: mITT
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3 | Cycle 4
Number analyzed (Participants) | 181 | 179 | 170 | 142
mm | -7.1 (23.8) | -3.3 (21.6) | -1.4 (15.4) | -1.5 (10.7)

ADVERSE EVENTS:
Time Frame: The visit schedule was comprised of six study visits: • Visit 1/Screening (4 weeks to 0 weeks prior to Visit 2) • Visit 2: (Day of/but prior to 1st chemotherapy treatment administration) • Visit 3: (Day of/but prior to 2nd chemotherapy treatment administration) • Visit 4: (Day of/but prior to 3rd, chemotherapy treatment administration) • Visit 5: (Day of/but prior to 4th, chemotherapy treatment administration) • Visit 6/Final Visit
Description: The safety population was equivalent to the modified intent to treat population (n=197) and included all patients who received at least one dose of the study treatment. Patients reported adverse events (excluding nausea and vomiting) in a diary from Day 1 to Day 5 post chemotherapy administration of each observation period. Safety events occurring between chemotherapy cycles were reported by the patient. Patients had a follow up period of 28 days post the last-chemotherapy cycle.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 9/197
Serious Adverse Events (participants affected / at risk) | 39/197
Other Adverse Events (participants affected / at risk) | 178/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=197)
Febrile Neutropenia (Blood and lymphatic system disorders) | 8 (10)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Metapneumovirus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Anal Ulcer (Gastrointestinal disorders) | 1 (1)
Diverticular Perforation (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Disease Progression (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Sudden Death (General disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Lower Gastrointestinal Haemorrhage (Vascular disorders) | 1 (1)
Septic Shock (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1)
Escherichia Bacteraemia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hallucination, Visual (Psychiatric disorders) | 1 (1)
Panic Attack (Psychiatric disorders) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Eosinophilic Cystitis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=197)
Fatigue (General disorders) | 89 (122)
Asthenia (General disorders) | 15 (17)
Decreased Appetite (General disorders) | 13 (13)
Constipation (Gastrointestinal disorders) | 58 (83)
Diarrhoea (Gastrointestinal disorders) | 35 (42)
Dyspepsia (Gastrointestinal disorders) | 34 (41)
Nausea (Gastrointestinal disorders) | 27 (32)
Abdominal Pain (Gastrointestinal disorders) | 11 (11)
Headache (Nervous system disorders) | 29 (38)
Dysgeusia (Nervous system disorders) | 14 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 46 (46)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 11 (19)
Neutropenia (Blood and lymphatic system disorders) | 16 (20)
Insomnia (Psychiatric disorders) | 11 (14)

LIMITATIONS AND CAVEATS:
The study was observational and open-label, lacking a control arm and randomization. Moreover, the study included mostly female patients and a high proportion of patients with breast or lung cancer, which may limit the generalizability of the study findings. Although "Quality of Life" data are subjective by nature, the FLIE questionnaire is validated, which minimizes the subjectivity of the patient-reported data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03649230/Prot_SAP_ICF_000.pdf